CLINICAL TRIAL: NCT02943460
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Subjects With Primary Sclerosing Cholangitis Without Cirrhosis
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of Cilofexor in Adults With Primary Sclerosing Cholangitis Without Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-428-4025; 2016-002442-23 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-10-24 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — cilofexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cilofexor 100 mg (Blinded Study Phase) (Experimental): Cilofexor 100 mg + placebo to match cilofexor 30 mg for up to 12.6 weeks
  Interventions: Drug: Cilofexor; Drug: Placebo to match cilofexor
- Cilofexor 30 mg (Blinded Study Phase) (Experimental): Cilofexor 30 mg + placebo to match cilofexor 100 mg for up to 12.7 weeks
  Interventions: Drug: Cilofexor; Drug: Placebo to match cilofexor
- Placebo (Blinded Study Phase) (Placebo Comparator): Placebo to match cilofexor 30 mg + placebo to match cilofexor 100 mg for up to 12.3 weeks
  Interventions: Drug: Placebo to match cilofexor
- Cilofexor (Open Label Extension Phase) (Experimental): Following the Blinded Study Phase, eligible participants received cilofexor for an additional up to 97.4 weeks.
  Interventions: Drug: Cilofexor

INTERVENTIONS:
Drug: Cilofexor — Tablet(s) administered orally once daily with food
  Other Names: GS-9674
  Arms: Cilofexor (Open Label Extension Phase); Cilofexor 100 mg (Blinded Study Phase); Cilofexor 30 mg (Blinded Study Phase)
Drug: Placebo to match cilofexor — Tablet(s) administered orally once daily with food
  Arms: Cilofexor 100 mg (Blinded Study Phase); Cilofexor 30 mg (Blinded Study Phase); Placebo (Blinded Study Phase)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of cilofexor in adults with primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PSC based on cholangiogram (magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP), or percutaneous transhepatic cholangiogram (PTC)) within the previous 12 months
* Serum alkaline phosphatase (ALP) > 1.67 x upper limit of the normal range (ULN)
* For individuals on ursodeoxycholic acid (UDCA), the dose of UDCA must have been stable for at least 12 months prior to screening through the end of treatment. For individuals not on UDCA, no UDCA use for at least 12 months before screening through the end of treatment
* For individuals being administered biologic treatments (eg, antitumor necrosis factor (TNF) or anti-integrin monoclonal antibodies), immunosuppressants or systemic corticosteroids, the dose must have been stable at least 3 months prior to screening and anticipated to remain stable throughout the trial
* Screening FibroSURE/FibroTest® <0.75 unless a historical liver biopsy within 12 months of screening does not reveal cirrhosis. In adults with Gilbert's syndrome or hemolysis, FibroSURE/FibroTest® will be calculated using direct bilirubin instead of total bilirubin.

Key Exclusion Criteria:

* Alanine aminotransferase (ALT) > 10 x ULN
* Total bilirubin > 2 x ULN
* International normalized ratio (INR) > 1.2 unless on anticoagulant therapy
* Small-duct PSC (histologic evidence of PSC with normal bile ducts on cholangiography)
* Other causes of liver disease including secondary sclerosing cholangitis and viral, metabolic, alcoholic, and other autoimmune conditions. Individuals with hepatic steatosis may be included if there is no evidence of nonalcoholic steatohepatitis (NASH) in the opinion of the investigator or on liver biopsy;
* Ascending cholangitis within 60 days of screening
* Presence of a percutaneous drain or bile duct stent
* Use of fibrates or obeticholic acid within 3 months prior to screening through the end of treatment
* Cirrhosis of the liver as defined by any of the following:

  * Historical liver biopsy demonstrating cirrhosis (eg, Ludwig stage 4 or Ishak stage ≥ 5)
  * Prior history of decompensated liver disease, including ascites, hepatic encephalopathy or variceal bleeding
  * Liver stiffness > 14.4 kilopascal (kPa) by FibroScan
* Current, active inflammatory bowel disease (IBD) defined as a partial Mayo score of > 1 and/or a score on the Rectal Bleeding domain > 0.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (23):
- United States (16):
  - University of California, Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Florida Digestive Health Specialists, Lakewood Rch, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Intermountain Medical Center - Transplant Services, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Universitätsklinik Klinik für Innere Medizin III, Vienna, Austria
- Canada (2):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - Toronto Liver Centre, Toronto, Ontario
- United Kingdom (4):
  - New Queen Elizabeth Hospital NHS Foundation Trust, Birmingham
  - Royal Free Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trauner M, Gulamhusein A, Hameed B, Caldwell S, Shiffman ML, Landis C, Eksteen B, Agarwal K, Muir A, Rushbrook S, Lu X, Xu J, Chuang JC, Billin AN, Li G, Chung C, Subramanian GM, Myers RP, Bowlus CL, Kowdley KV. The Nonsteroidal Farnesoid X Receptor Agonist Cilofexor (GS-9674) Improves Markers of Cholestasis and Liver Injury in Patients With Primary Sclerosing Cholangitis. Hepatology. 2019 Sep;70(3):788-801. doi: 10.1002/hep.30509. Epub 2019 Mar 10. PMID 30661255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 29 November 2016. The last study visit occurred on 18 May 2020.
Pre-assignment Details: 105 participants were screened.
Groups:
- Cilofexor 100 mg: Blinded Study Phase: Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily with food for up to 12.6 weeks
  Open Label Extension Phase: Cilofexor 100 mg tablet orally once daily with food for an additional up to 97.4 weeks
- Cilofexor 30 mg: Blinded Study Phase: Cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.7 weeks
  Open Label Extension Phase: Cilofexor 100 mg tablet orally once daily with food for an additional up to 97 weeks
- Placebo: Blinded Study Phase: Placebo to match cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.3 weeks
  Open Label Extension Phase: Cilofexor 100 mg tablet orally once daily with food for an additional up to 97 weeks
Period: Blinded Study Phase
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Started | 22 | 20 | 10
Completed | 19 | 19 | 10
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0
Period: Open Label Extension (OLE) Phase
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Started | 19 | 18 (1 participant completed the Blinded Study Phase, but did not continue in the OLE Phase.) | 10
Completed | 14 | 11 | 8
Not Completed | 5 | 7 | 2
Not completed — Adverse Event | 2 | 5 | 2
Not completed — Withdrew Consent | 2 | 1 | 0
Not completed — Investigator's Discretion | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Cilofexor 100 mg: Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily with food for up to 12.6 weeks
- Cilofexor 30 mg: Cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.7 weeks
- Placebo: Placebo to match cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.3 weeks
- Total: Total of all reporting groups
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 10 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.6) | 46 (12.1) | 42 (10.9) | 43 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 5 | 22
  Male | 11 | 14 | 5 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: Asian | 0 | 2 | 1 | 3
    Race: Black or African American | 4 | 3 | 1 | 8
    Race: White | 17 | 15 | 7 | 39
    Race: Not Permitted | 0 | 0 | 1 | 1
    Race: Other | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 0 | 3 | 0 | 3
    Ethnicity: Not Hispanic or Latino | 21 | 17 | 9 | 47
    Ethnicity: Not Permitted | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 2 | 2 | 8
  Austria | 1 | 0 | 0 | 1
  United States | 12 | 17 | 7 | 36
  United Kingdom | 5 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events During the Blinded Phase
Description: Treatment-emergent adverse events occurring during the Blinded Phase were defined as 1 or both of the following: 1) Any adverse events (AEs) with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug in the Blinded Phase (and before the first dosing date in the Open Label Extension (OLE) Phase), or 2) Any AEs leading to premature discontinuation of study drug in the Blinded Phase.
Time Frame: First dose date up to last dose date plus 30 days (Up to 17 weeks)
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 10
percentage of participants | 81.8 | 70.0 | 100.0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Serious Adverse Events During the Blinded Phase
Description: A serious adverse event was defined as an event that, at any dose, resulted in any of the following: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or a medically important event or reaction.
Time Frame: First dose date up to last dose date plus 30 days (Up to 17 weeks)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 10
percentage of participants | 13.6 | 0 | 0

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities During the Blinded Phase
Description: Treatment-emergent laboratory abnormalities occurring during the Blinded Phase were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug in the Blinded Phase plus 30 days (and prior to or on the first dose date of the OLE phase). The Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 was used for assigning toxicity grades (0 to 4, with higher grades indicating more severity).
Time Frame: First dose date up to last dose date plus 30 days (Up to 17 weeks)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 10
percentage of participants
  Any Grade 1 or Higher | 90.9 | 85.0 | 100.0
  Grade 1 | 22.7 | 25.0 | 10.0
  Grade 2 | 36.4 | 35.0 | 60.0
  Grade 3 | 27.3 | 20.0 | 30.0
  Grade 4 | 4.5 | 5.0 | 0

ADVERSE EVENTS:
Time Frame: Blinded Phase: First dose date up to last dose date plus 30 days (Up to 17 weeks); OLE Phase: First dose date up to last dose date plus 30 days (Up to 102 weeks)
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Cilofexor 100 mg (Blinded Phase): Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily with food for up to 12.6 weeks
- Cilofexor 30 mg (Blinded Phase): Cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.7 weeks
- Placebo (Blinded Phase): Placebo to match cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily with food for up to 12.3 weeks
- Cilofexor 100 mg (Open Label Extension Phase): Following the Blinded Phase, eligible participants received cilofexor 100 mg tablet orally once daily for an additional up to 97.4 weeks
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Cilofexor 30 mg (Blinded Phase) | Placebo (Blinded Phase) | Cilofexor 100 mg (Open Label Extension Phase)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/10 | 0/47
Serious Adverse Events (participants affected / at risk) | 3/22 | 0/20 | 0/10 | 10/47
Other Adverse Events (participants affected / at risk) | 18/22 | 14/20 | 10/10 | 41/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilofexor 100 mg (Blinded Phase) (N=22) | Cilofexor 30 mg (Blinded Phase) (N=20) | Placebo (Blinded Phase) (N=10) | Cilofexor 100 mg (Open Label Extension Phase) (N=47)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilofexor 100 mg (Blinded Phase) (N=22) | Cilofexor 30 mg (Blinded Phase) (N=20) | Placebo (Blinded Phase) (N=10) | Cilofexor 100 mg (Open Label Extension Phase) (N=47)
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 1 | 5
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 5
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pouchitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 1 | 0 | 2
Fatigue (General disorders) | 3 | 3 | 2 | 6
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 3
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 3
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 5 | 5 | 2 | 14
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 2
Viral infection (Infections and infestations) | 2 | 0 | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 2 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 4 | 2 | 7
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 3
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 6 | 20
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT02943460/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT02943460/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT02943460/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT02943460/Prot_003.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT02943460/SAP_004.pdf